CLINICAL TRIAL: NCT04127357
Title: Progression of Active Microcavitated Carious Lesions on Primary Teeth Occlusal Surfaces: Randomize Clinical Trial
Brief Title: Progression of Active Microcavitated Carious Lesions on Primary Molar Occlusal Surfaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, PhD, Senior Lecturer, Clinical Professor, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLM 8
Record Dates: First submitted 2019-08-12; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Dental Caries in Children; Pit and Fissure Sealant; Toothbrushing
Keywords: Pit and fissure sealants; Pediatric dentistry; Toothbrushing
MeSH Terms: conditions — Van der Woude syndrome | interventions — CMW cement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Control (Other): Brushing with 1450 ppm fluoride toothpaste.
  Interventions: Procedure: 1450 ppm fluoride toothpaste brushing x Resin sealing (FluroShield, Dentsply, Brazil).
- B - Test (Experimental): Resin sealing (FluroShield, Dentsply, Brazil).
  Interventions: Procedure: 1450 ppm fluoride toothpaste brushing x Resin sealing (FluroShield, Dentsply, Brazil).

INTERVENTIONS:
Procedure: 1450 ppm fluoride toothpaste brushing x Resin sealing (FluroShield, Dentsply, Brazil). — After randomization of the children, the selected molars were allocated through a randomized sequence list in 2 groups: A. Brushing with 1450 ppm fluoride toothpaste, donated by the researcher; B. Resin Sealing (FluroShield, Dentsply, Brazil).
  The teeth included in the second group (group B) underwent a second randomization: B1. With absolute isolation; B2. With relative isolation. For the group with absolute isolation, topical anesthesia and local papillary infiltration were performed for subsequent staple placement. Relative isolation was performed with cotton rollers and moisture control suction. The sealant selected was the opaque fluroshield to facilitate visualization upon visual examination during reevaluations and was applied following the manufacturer's standards. The teeth were clinically and radiographically followed at 6 and 12 months and two sessions of motivation reinforcement were performed through video and brush change at 3 and 9 months.

SUMMARY:
Objective: To verify the progression of active microcavitated carious lesions on occlusal surfaces of primary molars after the orientation of the brushing technique associated with fluoride dentifrice compared to resin sealant, through a 12-month randomized clinical trial. Methodology: We selected 22 children from 4 to 9 years old from the public school system of the city of Juazeiro do Norte-Ceará, with at least one primary molar presenting an active caries lesion score 3 of the International Caries Detection and Assessment System (ICDAS). Randomization was performed en bloc and stratified by two conditions (age and caries experience). The selected teeth were divided into two groups: the first (G1) was submitted to brushing with fluoridated toothpaste; and the other group (G2) to the resin sealing technique, whose application of the material was performed under absolute or relative isolation, selected through a second randomization. The molars undergoing treatment were evaluated at 6- and 12-month returns. Caries progression was evaluated according to the type of treatment, dental group and sealant retention by the Chi-square test. For cost analysis, the variance test (ANOVA) was used.

ELIGIBILITY:
Inclusion Criteria:

* At least one primary molar with active caries lesions classified as ICDAS score 3.

Exclusion Criteria:

* Children with differentiated management needs and/or systemic diseases with oral involvement.
* Primary molar with active caries lesions classified as ICDAS score 3 that had other caries lesions involving dentin, restorations, sealants, or other types of formation defects.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of caries progression | 6 months
  With the radiographs in hand, the possible progression of the treated caries lesion was observed, which was coded as: a) Absent progression: no radiolucent area of the lesion; b) Present progression: with increase in the radiolucent area of the lesion.
Clinical evaluation of caries progression | 12 months
  With the radiographs in hand, the possible progression of the treated caries lesion was observed, which was coded as: a) Absent progression: no radiolucent area of the lesion; b) Present progression: with increase in the radiolucent area of the lesion.

SECONDARY OUTCOMES:
Sealant retention | 6 months
  Clinical evaluation of sealant retention was performed using the criteria used by Pardi: RT- total retention, PP1- presence of sealant on two thirds of the occlusal surface, PP2- presence of sealant on one third of the occlusal surface. PT-total loss of sealant on occlusal surface.
Sealant retention | 12 months
  Clinical evaluation of sealant retention was performed using the criteria used by Pardi: RT- total retention, PP1- presence of sealant on two thirds of the occlusal surface, PP2- presence of sealant on one third of the occlusal surface. PT-total loss of sealant on occlusal surface.

OTHER OUTCOMES:
Direct cost estimate | 6 months
  To estimate costs, the sessions were timed (initial and reevaluations) and for each consultation a table was filled in, which should contain the quantities of materials used per session. Prices of materials were considered by inferring the market value obtained by an average of 3 (three) different places that market the products in question, thus obtaining different costs for the proposed treatments.
Direct cost estimate | 12 months
  To estimate costs, the sessions were timed (initial and reevaluations) and for each consultation a table was filled in, which should contain the quantities of materials used per session. Prices of materials were considered by inferring the market value obtained by an average of 3 (three) different places that market the products in question, thus obtaining different costs for the proposed treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carlos P Imparato, PhD, Principal Investigator — Sao Leopoldo Mandic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meyer-Lueckel H, Paris S. When and How to Intervene in the Caries Process. Oper Dent. 2016 Sep;41(S7):S35-S47. doi: 10.2341/15-022-O. PMID 27689929
- [Result] Bakhshandeh A, Qvist V, Ekstrand KR. Sealing occlusal caries lesions in adults referred for restorative treatment: 2-3 years of follow-up. Clin Oral Investig. 2012 Apr;16(2):521-9. doi: 10.1007/s00784-011-0549-4. Epub 2011 Apr 9. PMID 21479565